CLINICAL TRIAL: NCT02543866
Title: Fecal Microbiota Transplantation as a Strategy to Eradicate Intestinal Carriage of Resistant Organisms
Brief Title: Fecal Microbiota Transplantation as a Strategy to Eradicate Resistant Organisms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Danielle Zerr, Professor, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15587
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Infection Resistant to Drugs
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Subjects will receive 50mL of prepared stool fecal via nasogastric tube
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation

SUMMARY:
This protocol will evaluate fecal microbiota transplantation (FMT) as a strategy to eradicate intestinal colonization of extended-spectrum resistant (ESC-R) Enterobacteriaceae in pediatric patients.

FMT will be performed on subjects with a history of at least one infection due to ESC-R Enterobacteriaceae.

This protocol aims to determine the feasibility, safety, tolerability, and potential efficacy of FMT in pediatric patients with a history of ESC-R Enterobacteriaceae.

DETAILED DESCRIPTION:
This is a prospective pilot study of fecal microbiota transplantation in pediatric patients with a history of ESC-R Enterobacteriaceae. Subjects who meet inclusion/exclusion criteria and provide written, informed consent will undergo screening studies and provide a pre-FMT stool sample to confirm intestinal carriage of ESC-R Enterobacteriaceae. The FMT will be administered by nasogastric tube in the outpatient setting by trained personnel. The subjects will be monitored for potential adverse events, recurrence of MDRO infections, infections that may be related to FMT, and worsening of existing comorbidities or development of new comorbidities for the 12 months post-FMT with the option of participating in long-term follow-up for up to 5 years post-FMT. Patients will provide stool samples 2 days, 2 weeks, 4 weeks, 8 weeks, 6 months, and 12 months post-FMT. These samples will be testing for ESC-R Enterobacteriaceae.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents between 7 and 21 years of age.
2. A history at least one infection due to ESC-R Enterobacteriaceae. ESC-R isolates will be defined as those non-susceptible to ceftriaxone, cefotaxime, or ceftazidime.
3. Parent/guardian and participant must be able to attend baseline and follow-up study visits.
4. Subject must be willing and able to provide written informed consent or assent (as appropriate by age).

Exclusion Criteria:

1. Patients with any history of malignancy or any immunocompromised state (e.g. absolute neutrophil count outside the normal range) induced by disease or therapy will be excluded.
2. Patients with past or current use of systemic immunosuppressive agents will be excluded. Receipt of non-systemic agents such as inhaled, nasal, or topical steroids or immune-modulating agents are allowed.
3. Lack of intestinal carriage of ESC-R Enterobacteriaceae (negative selective stool culture for ESC-R Enterobacteriaceae).
4. Allergy or hypersensitivity to omeprazole and polyethylene glycol.
5. Pregnancy.
6. Current history of frequent (>1 per week) vomiting.
7. Active inflammatory gastrointestinal disease, such as inflammatory bowel disease
8. Active mucositis or acute graft versus host disease of the gastrointestinal tract
9. Concurrent abdominal radiation therapy.
10. Inability to tolerate nasogastric tube placement or contraindication to having an NG tube placed.
11. Presence of a ventriculoperitoneal shunt or other intrabdominal device, receipt of renal dialysis, presence of ascites, or other conditions/devices that would increase the risk of peritonitis.
12. Bleeding diatheses
13. Patients with current active ESC-R Enterobacteriaceae infection who have not yet completed antibiotic treatment will be excluded until their treatment is completed

    -

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of FMT as measured by Incidence, severity, and relatedness of solicited, unsolicited, and serious adverse events | 12 months post-FMT; optional long-tern follow-up for 5 years post-FMT
  Incidence, severity, and relatedness of solicited, unsolicited, and serious adverse events

SECONDARY OUTCOMES:
Efficacy of FMT | 2 days, 2 weeks, 4 weeks, 8 weeks, 6 months, 12 months post-FMT
  Proportion of subjects free from ESC-R intestinal colonization and recurrent ESC-R infections 2 days, 2 weeks, 4 weeks, 8 weeks, 6 months, and 12 months post-FMT

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Zerr, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No